CLINICAL TRIAL: NCT06930170
Title: Evaluation of Cochlear Implantation in Unilateral or Asymmetric Hearing Loss in Children.
Acronym: AsymIC-Ped
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220669; 2023-A00003-42 (Other: ID-RCB Number)
Record Dates: First submitted 2025-03-31; First posted 2025-04-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Unilateral Hearing Loss; Asymmetric Hearing Loss
Keywords: Cochlear implants; unilateral hearing loss; Asymmetric hearing loss
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cochlear implant (Experimental): Fitted with a cochlear implant
  Interventions: Device: CROS or BiCROS device fitting; Diagnostic Test: French simplified matrix test (FraSimat); Diagnostic Test: Sound localization test (ERKI); Diagnostic Test: Cortical Auditory Evoked Potentials (PEAc); Other: Speech, Spatial and Qualities of Hearing Scale (SSQ); Other: Peabody Picture Vocabulary Scale (PPVT or EVIP in french); Other: NEPSY-II (A Developmental Neuropsychological Assessment); Other: Pediatric Quality of Life Inventory™ Multidimensional Fatigue Scale (PedsQL MFS)
- CROS or biCROS system (Active Comparator): Fitted with a CROS or BiCROS system, depending on the type of hearing loss
  Interventions: Device: Cochlear implantation; Diagnostic Test: French simplified matrix test (FraSimat); Diagnostic Test: Sound localization test (ERKI); Diagnostic Test: Cortical Auditory Evoked Potentials (PEAc); Other: Speech, Spatial and Qualities of Hearing Scale (SSQ); Other: Peabody Picture Vocabulary Scale (PPVT or EVIP in french); Other: NEPSY-II (A Developmental Neuropsychological Assessment); Other: Pediatric Quality of Life Inventory™ Multidimensional Fatigue Scale (PedsQL MFS)

INTERVENTIONS:
Device: Cochlear implantation — During surgery at 8 weeks after inclusion, cochlear implant is implanted
  Arms: CROS or biCROS system
Device: CROS or BiCROS device fitting — At 8 weeks after inclusion, CROS or BICROS (depending on the type of hearing loss) is fitting
  Arms: Cochlear implant
Diagnostic Test: French simplified matrix test (FraSimat) — The FraSimat is an adaptive test that measures speech intelligibility in noise. It consists of 14 sentences of 3 words each, recorded in the presence of background noise. The FraSimat will be performed in two different configurations in relation to the source of the signal and noise before implantation or fitting, and 1, 2, 3 and 4 months after.
Diagnostic Test: Sound localization test (ERKI) — ERKI for German "Erfassung des Richtungshörens für Kinder" is an automated test that assesses spatial localization skills. The test is performed with the child seated facing a semi-circular table, surrounded by a set of 5 loudspeakers arranged 1 meter apart.
  The test consists of 5 stimuli, followed by 42 trials. Following the presentation of each stimulus, the child must turn a control knob and direct the LED light to the point where he or she has perceived it. The child validates his or her response by pressing the button.
  ERKI is evaluated before implantation or fitting, and 1, 2 and 3 months after.
Diagnostic Test: Cortical Auditory Evoked Potentials (PEAc) — The recording of Auditory Cortical Evoked Potentials provides an objective means of assessing the maturation of the auditory system and its ability to process auditory signals. AEPs consist of a series of cortical responses to an auditory stimulus.
  PEAc are assessed using a non-invasive EEG recording, made under quiet wakefulness. Four surface electrodes are glued to the patient's skull: one on the vertex, one on the forehead, and one on each mastoid. The latency (msec) and amplitude (mV) values of each of the four component waves will be analyzed.
  PEAc is evaluated before implantation or fitting, and 3 and 4 months after.
Other: Speech, Spatial and Qualities of Hearing Scale (SSQ) — The Speech, Spatial and Qualities of Hearing Scale is a questionnaire for subjective evaluation of listening performance in everyday listening situations. The parent version is adapted for parents of hearing-impaired children.
  SSQ is evaluated before implantation or fitting, and 4 months after.
Other: Peabody Picture Vocabulary Scale (PPVT or EVIP in french) — Peabody Picture Vocabulary Scale assesses the extent of French listening vocabulary acquired by the child.
  The PPVT is designed for patients aged from 2 years and 6 months to 18 years. The raw score is the number of images correctly identified.
  Peabody Picture Vocabulary Scale is evaluated before implantation or fitting, and 4 months after.
Other: NEPSY-II (A Developmental Neuropsychological Assessment) — The NEPSY-II (A Developmental Neuropsychological Assessment) is a battery of neuropsychological tests designed to assess children's skills in 6 major neuropsychological domains. The various tests are validated for the age range indicated in brackets, and will be used for patients aged 5 and over.
  NEPSY-II is evaluated before implantation or fitting, and 4 months after.
Other: Pediatric Quality of Life Inventory™ Multidimensional Fatigue Scale (PedsQL MFS) — PedsQL MFS is a questionnaire used to assess subjective experiences of fatigue. The questionnaire consists of 18 items The parent version is adapted for parents of hearing-impaired children. PedsQL MFS is evaluated before implantation or fitting, and 4 months after.

SUMMARY:
Today, unilateral hearing loss must be assessed and managed just as bilateral hearing loss is. It is recommended to consider the auditory difficulties caused by the loss of stereophonic hearing and to offer auditory rehabilitation as early as possible. Studies show that hearing devices can be effective in certain cases and for specific auditory modalities. The prognostic factors for successful hearing aid adaptation are linked to early intervention and the presence of residual hearing (using a BiCROS system). However, the cochlear implant remains the only device capable of potentially restoring contralateral auditory function in cases of single-sided deafness (SSD) and severe to profound unilateral hearing loss with asymmetrical deafness

DETAILED DESCRIPTION:
Unilateral congenital deafness has significant repercussions on a child's development. Numerous studies on this population have demonstrated its impact on speech and language development, as well as academic progress. Monaural hearing increases the risk of listening fatigue and causes considerable difficulty in sound localization and speech perception in noisy environments, as these abilities rely on binaural hearing.

Recent research has also indicated that in children with unilateral deafness, the better ear may be affected by sensory deprivation in the impaired ear. Despite these substantial effects, treatment options for these children remain limited. Traditional hearing aids are insufficient to restore functional hearing in cases of profound deafness. The only routinely available options are a Bone-Anchored Hearing Aid (BAHA) or a Contralateral Routing of Sound (CROS) system. While these devices allow the signal from the affected side to be transmitted to the better ear, they do not restore binaural hearing, unlike cochlear implants (CIs).

A growing body of evidence has demonstrated the benefits of cochlear implantation on speech perception in noise and sound localization in adults. However, in France, CIs are currently indicated only for cases of severe to profound unilateral deafness associated with debilitating tinnitus, and only when alternative treatments-such as CROS systems and osseointegrated hearing aids-have failed in children. While studies suggest that children may achieve similar outcomes, no clinical research has been conducted. This study aims to evaluate functional performance and neurological correlates in unilaterally implanted children with unilateral hearing loss, in comparison with their hearing-aided peers

ELIGIBILITY:
Inclusion Criteria:

* Child aged 4 to 6 years at the time of inclusion
* Using spoken French as the primary mode of communication
* Diagnosed with unilateral or asymmetric hearing loss :

Unilateral is defined by severe to profound hearing loss in the affected ear (thresholds > 70 dB at ≥ 4 frequencies, established by audiometry or ASSR) and normal hearing in the better ear (thresholds ≤ 25 dB between 500-4000 Hz, established by audiometry or ASSR).

Asymmetric is defined by severe to profound hearing loss in the weaker ear (thresholds > 70 dB at ≥ 4 frequencies, established by audiometry or ASSR) and mild hearing loss in the better ear (thresholds between 30-40 dB at ≤ 4 frequencies, established by audiometry or ASSR).

* Written informed consent from both legal guardians (or the sole guardian, if applicable)
* Affiliated with a health insurance system or entitled to coverage

Exclusion Criteria:

* Severe neurological disorder, identified by MRI and/or a neuro-pediatric assessment
* Severe cognitive, child psychiatric, or developmental delay
* Severe cochleo-vestibular malformation
* Severe cochlear nerve malformation
* Social circumstances preventing long-term follow-up
* Family not proficient in spoken French
* Patient fitted with a CROS or BiCROS system
* Patient with a contraindication to implantation surgery or anesthesia (including lack of meningitis/pneumococcal vaccination)

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
French simplified matrix test (FraSimat) SAABAN condition at Month 18 | 18 months after implantation or fitting
  The primary endpoint is intervention success, defined as an increase ≥ 6dB SNR (Signal-to-Noise Ratio) at 18 months compared with the value at the pre-intervention visit. It is assessed in the SAABAN condition, i.e. by presenting the signal (speech) to the better ear and the noise to the better ear.

SECONDARY OUTCOMES:
French simplified matrix test (FraSimat) SAABAN condition at Month 12 | 12 months after implantation or fitting
  Evolution of FraSimat score in Signal to Noise Ratio at 12 months compared with the value at the pre-intervention visit. It is assessed in the SAABAN condition, i.e. by presenting the signal (speech) to the better ear and the noise to the better ear.
French simplified matrix test (FraSimat) S0B0 condition at Month 18 | 18 months after implantation or fitting
  Evolution of FraSimat score in Signal to Noise Ratio at 18 months compared with the value at the pre-intervention visit. It is assessed in the S0B0 condition, i.e. signal and noise at 0° to the head (in front).
French simplified matrix test (FraSimat) S0B0 condition at Month 12 | 12 months after implantation or fitting
  Evolution of FraSimat score in Signal to Noise Ratio at 12 months compared with the value at the pre-intervention visit. It is assessed in the S0B0 condition, i.e. signal and noise at 0° to the head (in front).
Sound localization test (ERKI) Month 12 | 12 months after implantation or fitting
  Evolution of RMSE (root-mean-square deviation) in the ERKI (Assessment of directional hearing for children) test between the pre-intervention visit and Month 12
Sound localization test (ERKI) Month 18 | 18 months after implantation or fitting
  Evolution of RMSE (root-mean-square deviation) in the ERKI (Assessment of directional hearing for children) test between the pre-intervention visit and Month18
Questionnaire Speech, Spatial and Qualities of Hearing Scale (SSQ, version parent) | 18 months after implantation or fitting
  Evolution of SSQ total score and sub-scores between the pre-intervention visit and Month 18.
Peabody Picture Vocabulary Scale (PPVT or EVIP in french) | 18 months after implantation or fitting
  Change in standardized PPVT/EVIP score from pre-intervention visit to Month 18
NEuroPSYchological assessment NEPSY-II | 18 months after implantation or fitting
  Change in NEPSY-II score between pre-intervention visit and Month 18 in patients aged 5 and over at inclusion.
Cortical Auditory Evoked Potentials (PEAc) Month 12 | 12 months after implantation or fitting
  Evolution of latencies and amplitudes between the pre-intervention visit and Month12 for waves P1, N1, P2, N2.
  Evolution of the interaural difference in P1 latency between the pre-intervention visit and Month 12 (experimental group only).
Cortical Auditory Evoked Potentials (PEAc) Month 18 | 18 months after implantation or fitting
  Evolution of latencies and amplitudes between the pre-intervention visit and Month18 for waves P1, N1, P2, N2.
  Evolution of the interaural difference in P1 latency between the pre-intervention visit and Month 18 (experimental group only).
Quality of life : Pediatric Quality of Life Inventory Multidimensional Fatigue Scale (PedsQL MFS) | 18 months after implantation or fitting
  Evolution of the PedsQL MFS total score and sub-scores between the pre-intervention visit and Month18.
Device satisfaction | Up to 18 months after implantation or fitting
  Duration of device use via datalogging of implant cochlear or hearing system
Number of adverse events | Up to 18 months after implantation or fitting
  Expected implant-related adverse events may include Facial paralysis or paresis, Dizziness, Meningitis, Skin complications, Implant failure The presence of one or more of these effects will be evaluated at each ENT (ear nose throat) assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LOUNDON, MD, PHD, Study Chair — Unité d'Audiophonologie et d'Implantation cochléaire - Service d'ORL et chirurgie cervico-faciale Hôpital Necker.
Locations (1):
- Audiophonology Unit of the Ear, Nose and Throat (ENT) Department ("Oto-rhino-laryngologie (ORL) et chirurgie cervico-faciale"), Paris, France

IPD SHARING:
Plan to Share IPD: No